CLINICAL TRIAL: NCT06245707
Title: To Evaluate the Effects of Different Treatment Schemes on Cognitive Function of Patients With Idiopathic Membranous Nephropathy and Explore the Possible Mechanism by Using Functional Magnetic Resonance Imaging (fMRI)
Brief Title: the Effects of Different Treatment Schemes on Cognitive Function of Patients With Idiopathic Membranous Nephropathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-P2-233
Record Dates: First submitted 2023-09-25; First posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2023-09

CONDITIONS: Mild Cognitive Impairment; Idiopathic Membranous Nephropathy
MeSH Terms: conditions — Cognitive Dysfunction; Glomerulonephritis, Membranous | interventions — Prednisone; Cyclophosphamide; Rituximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ponticelli group (Experimental): Patients with idiopathic membranous nephropathy were treated with Ponticelli protocol,that is alternating prednisone or methylprednisone -cyclophosphamide every other month
  Interventions: Drug: prednisone,methylprednisone and cyclophosphamide
- Rituximab group (Experimental): Patients with idiopathic membranous nephropathy were treated with Rituximab.The specific dosage of rituximab depends on the guidance of peripheral blood B cells.
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: prednisone,methylprednisone and cyclophosphamide — In the first month, methylprednisolone 500mg/d was given intravenously for 3 days, and then prednisone 0.5 mg/(kg d) * for 27 days. Oral cyclophosphamide 2.0 mg/(kg d) * 30 days in the second month. After that, the first month and the second month plan were repeated twice.
  Arms: Ponticelli group
Drug: Rituximab — The dosage of rituximab depends on peripheral blood B cells. After the treatment of rituximab, the peripheral blood B cells were in a clear state and then stopped. After monitoring the recovery of B cells, additional doses were given.
  Arms: Rituximab group

SUMMARY:
This study intends to apply prospective, open, single-center, randomized controlled study to evaluate the cognitive status of patients with Idiopathic membranous nephropathy and the influence of different treatment schemes on the cognitive status of patients with Idiopathic membranous nephropathy, and explore the possible pathophysiological mechanism by using brain magnetic resonance imaging technology.

DETAILED DESCRIPTION:
Proteinuia is an independent risk factor for cognitive dysfunction and dementia. There is no relevant research on whether patients with Idiopathic membranous nephropathy with normal renal function are complicated with cognitive impairment. In the process of clinical diagnosis and treatment, it was observed that the cognitive function of patients with Idiopathic membranous nephropathy decreased significantly after treatment compared with that before treatment. However, there is no clinical study to confirm this phenomenon at present, and the causes of cognitive function damage are not clear. This study intends to apply prospective, open, single-center, randomized controlled study to evaluate the cognitive status of patients with Idiopathic membranous nephropathy and the influence of different treatment schemes on the cognitive status of patients with Idiopathic membranous nephropathy, and explore the possible pathophysiological mechanism by using brain magnetic resonance imaging technology, so as to fill the research gap of clinical cognitive status of Idiopathic membranous nephropathy and provide theoretical basis for better clinical treatment scheme selection and prevention of cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with nephrotic syndrome and normal renal function.
* Patients with idiopathic membranous nephropathy diagnosed by pathology.
* not received hormone or other immunosuppressive treatment in the past six months.

Exclusion Criteria:

* Unable to treat patients with hormones and immunosuppression.
* Patients with definite intracranial diseases such as previous cerebral infarction and cerebral hemorrhage;
* Patients who have been diagnosed with cognitive decline or dementia in the past;
* Patients with claustrophobia or have other contraindications for magnetic resonance imaging, such as pacemakers and metal foreign bodies in the body.
* Pregnant and lactating women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
The cognitive function of the two groups was evaluated and analyzed by the Chinese version of Montreal Cognitive Assessment Scale (MoCA) | enrollment, half a year after treatment and one year after treatment.
  The two groups of patients were given a quiet environment and completed the test within 10 minutes. The cognitive function of the two groups was evaluated and analyzed by the Chinese version of Montreal Cognitive Assessment Scale (MoCA). The possible score was between 0 and 30. The higher the score, the better the cognitive state. We defined cognitive impairment as a total score of less than 26 for participants with high school education or below and less than 27 for participants with high school education or above, because the average score of MOCA varies according to the level of education

SECONDARY OUTCOMES:
Brain magnetic resonance high-resolution structural imaging was performed to observe the changes of brain structure | enrollment, half a year after treatment and one year after treatment.
  All participants were examined with 3.0T MRI scanner (GE Healthcare, discovery mr750w, Milwaukee, WI), using quantitative techniques such as high-resolution structural magnetic resonance, resting state functional magnetic resonance and arteriovenous spin labeling imaging (ASL).

CONTACTS AND LOCATIONS:
Overall Officials: Jia Wang, Principal Investigator — Student
Locations (1):
- Beijing Friedship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No